CLINICAL TRIAL: NCT06067009
Title: A Feasibility Trial of a Stakeholder-Enhanced, Lay-Navigator-Delivered Intervention to Improve the Decisional Partnership of Chronic Kidney Disease Dyads
Brief Title: Feasibility Trial of a Stakeholder-enhanced Lay-navigator-delivered Intervention (ImPart-Multi)
Acronym: ImPart-Multi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Shena Gazaway, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 300011311; UAB (Other Grant/Funding Number: Forge AHEAD)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Kidney Diseases; Cardiometabolic Risk Factors
Keywords: decision support; decision-making; patient activation; caregiving
MeSH Terms: conditions — Kidney Diseases; Patient Participation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 - Communication (Experimental): Participants in this group will complete one session of communication training and will have 1 follow up call a month after the session has been completed.
  Interventions: Behavioral: ImPart-Multi - IMproving the decisional PARTnership of Chronic Kidney Disease Dyads with concurrent metabolic disease
- Group 2 - Social Support Effectiveness (Experimental): Participants in this group will complete 3 sessions of social support effectiveness training. All will complete 1 follow-up call after the 3 sessions have been completed.
  Interventions: Behavioral: ImPart-Multi - IMproving the decisional PARTnership of Chronic Kidney Disease Dyads with concurrent metabolic disease
- Group 3 - Communication and Social Support Effectiveness (Experimental): Participants assigned to this group will complete 4 sessions of communication and social support effectiveness training. One follow up call will be completed one month after the last session has been competed.
  Interventions: Behavioral: ImPart-Multi - IMproving the decisional PARTnership of Chronic Kidney Disease Dyads with concurrent metabolic disease
- Group 4 - Wait-listed Control (Placebo Comparator): Participants assigned to this group will receive no training sessions the first 12 weeks of enrollment. After 12 week data collection, they will be assigned to complete either communication (1 session) or social support effectiveness (3 sessions) training. One month after the completion of the training sessions a follow-up call will be made.
  Interventions: Behavioral: ImPart-Multi - IMproving the decisional PARTnership of Chronic Kidney Disease Dyads with concurrent metabolic disease

INTERVENTIONS:
Behavioral: ImPart-Multi - IMproving the decisional PARTnership of Chronic Kidney Disease Dyads with concurrent metabolic disease — ImPart-Multi is a psychoeducational, decision support training program, designed to impact Black chronic kidney disease patients with concurrent metabolic disease and their care partners' ability to 1. contemplate the decision needed, 2. request resources/support, and 3. make an informed patient-centered decision. Participants will participate in either communication training, social support effectiveness training, or a combination of both.

SUMMARY:
We seek to explore the feasibility and acceptability of participation in a decision-support training program led by lay navigators. ImPart-Multi, an education-telehealth-based, is designed to empower Black chronic kidney disease patients (CKD) patients and their care partner to seek the resources and support needed to be activated allies when making health-related decisions.

Participants, based on random assignment, will participate in survey completion at study start and at 12 and 24 weeks of enrollment, and will complete 1, 3, or 4 education sessions via telehealth or audio connection. Participants will also complete an interview to share their thoughts on the program and other factors of interest.

DETAILED DESCRIPTION:
Black people with chronic kidney disease and uncontrolled high blood pressure face a higher risk of developing severe cardiovascular disease and face an additional risk of their kidney disease getting worse more quickly. Many things add to this risk, including living in areas with lower access to support resources and lower quality of communication and information sharing with medical team members. Over the past 18 months, our team has worked in partnership with a group of community advisory members, two who are living with chronic kidney disease, two who are care partners of someone with chronic kidney disease, and one who has experience as a social worker in a dialysis clinic. Together we have created a program focused on teaching skills for health-related decision-making. The program consists of education on 1) communication, 2) social support usefulness, or 3) a combination of both. We seek to understand how these sessions, alone or together, impact how the person with chronic kidney disease makes decisions and how they feel they receive support from their care partner and/or medical team. We also seek to understand if there are benefits to the person with chronic kidney disease and their care partner's quality of life and how the two work together to cope with the illness experience. Our goal is to positively impact health promotion by teaching answer-seeking behaviors to people with high-risk chronic kidney disease.

Our team will recruit 32 Black adults with stage 3 or 4 chronic kidney disease and one identified care partner for a total of 64 people from the University of Alabama at Birmingham (UAB) Chronic Kidney Disease Clinic and Cooper Green Primary and Kidney Specialty Care Clinic. In the study, there are four groups of participants: Group 1 will participate in one session on communication, Group 2 will receive 3 sessions on social support effectiveness; and Group 3 will have both communication and social support sessions. Group 4 will not participate in the sessions at all. All groups will be asked to complete surveys and one interview about their experience three months after the program is done. After this data collection, the participants in Group 4 will be invited to participate in the session combination they choose, so they receive potential benefit from their participation.

Participants will be paid $20 when they complete surveys at three points - 1) when starting the study, 2) at the end of three months, and 3) if the participant completes the interview. The education sessions will be delivered over video conference connection with those lacking access or the ability to connect using audio only.

We plan to share our results scientifically and in the community as a team. Our plans for community sharing is through group classes, developed from content that was shared as beneficial in the interviews at Cooper Green and the UAB Chronic Kidney Disease Clinic and in two community-based locations that the community advisory group identifies. Our team, including our community advisory croup members, will also write articles to submit to science-based journals. The results of this project will be used to prepare and submit an application to receive more funding to evaluate this program with a larger group of people from other areas in the state or the country.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  1. Electronic medical record (EMR) documented diagnosis of stage 3 or 4 CKD (2 estimated glomerular filtration rate [eGFR] between 45-15 within 90 days); and concurrent cardiometabolic disease (hypertension and/or diabetes)
  2. Ability to speak and read English and complete baseline questionnaires;
  3. Patients must have a care partner enrolled in the study - the team will assist any patient in identifying a care partner, if interested.

Inclusion Criteria:

* Care partner

  1. Age ≥18; 2) Self-endorsing or identified by the patient as "a relative, friend, or partner that has a close relationship with you and who assists you with your medical decisions and who may or may not live in the same residence as you and who is not paid for their help";
  2. Ability to speak and read English and complete baseline questionnaires;
  3. Care partners must have an enrolled patient.

Exclusion Criteria:

* Patients

  1. Receiving hospice;
  2. Receiving dialysis;
  3. Medical record documentation of active unmedicated severe mental illness, moderate-severe dementia, suicidal ideation, uncorrected hearing loss, and active substance abuse.

Exclusion Criteria:

* Care partner 1. Self-reported unmedicated mental illness, mild-severe dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse ascertained by study introduction questioning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention and Study Procedures | Baseline to 12 weeks Groups 1, 2 and 3; 24 weeks Group 4
  Through qualitative interviews, participant reported experiences with the ImPart Multi intervention and trial procedures.
Feasibility of Intervention Delivery and Data Collection | Groups 1, 2, 3 and 4 baseline through to 12 weeks; Group 4 only baseline to 24 weeks
  Proportion of participants who complete assigned intervention group and study related assessments.

SECONDARY OUTCOMES:
Decision-making process using the Decision Conflict Scale (DCS) | baseline, and 24 weeks after baseline
  16 items total; measures perceptions of uncertainty in choosing options, factors contributing to uncertainty and feeling that decisions were informed and values-based
Decision-making process using the Social Support Effectiveness-Questionnaire | baseline and 12 weeks after baseline
  25 items measuring perceptions of help received in last 3 months
Patient Wellbeing using the Kidney Disease Quality of Life Scale (KDQOL-36) | baseline and 12 weeks after baseline
  36 items measure 3 components:physical health, mental health, and kidney disease health.
Care partner well being using the PROMIS Global Health 10 | baseline and 12 weeks after baseline
  10 items measure global health-related quality of life in 2 domains, physical and mental health
Dyadic Interaction using the Dyadic Coping Inventory | baseline and 12 weeks after baseline
  37 item instrument designed to measure perceived communication and dyadic coping in close relationships when one or both partners is stressed.

CONTACTS AND LOCATIONS:
Overall Officials: Shena Gazaway, PhD, Principal Investigator — UAB School of Nursing
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No